CLINICAL TRIAL: NCT03417817
Title: Measurement of Acid Exposure in Healthy Subjects Using 96 Hours Wireless pH Monitoring (Bravo™)
Brief Title: Oesophageal Acid Exposure in Healthy Subjects Over 96 Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 227671
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: healthy subjects and subjects referred for gastroscopy in context of other conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects (Other): Bravo wireless pH monitoring over 96 hours
  Interventions: Device: Bravo

INTERVENTIONS:
Device: Bravo — wireless pH monitoring over 96 hours

SUMMARY:
First introduced over 40 years ago, the 24-hour catheter-based pH studies have previously been found to be the gold standard in the diagnosis of gastro-oesophageal reflux disease (GORD). In 2003, the Bravo has revolutionised the study of GORD, allowing patients an improved comfort and ability to perform activities of daily living.

The backflow of gastric acid (acid exposure) in the oesophagus is monitored by a tiny pH sensor located in a capsule which is pinned temporarily to the wall of the oesophagus at the time of endoscopy. Normal measurements for acid exposure are established for 48-hour studies. However, the investigators' studies have shown that extending the duration of recording to 96 hours further improved the diagnostic yield for GORD in patients with negative 24-hour catheter-based tests

The 96-hour recording is the current standard of care, despite the lack of normal ranges for this duration of the recording. The basis for the diagnosis of GORD in 96-hours studies is based on the 48-hours normal controls. The objective of this study is to determine the normal values for oesophageal acid exposure using the wireless pH recording apparatus over 96 hours in asymptomatic healthy subjects with unrestricted activity and diet.

DETAILED DESCRIPTION:
This is a single centre study on healthy subjects to determine the normal values for oesophageal acid exposure using the wireless pH monitoring over 96 hours. The investigators anticipate the recruitment of 50 participants over 10 months.

Subjects without reflux symptoms, either healthy volunteers (hospital staff and medical students) or people referred for gastroscopy in the context of other conditions (e.g. iron deficiency anaemia, suspected coeliac disease) will be recruited. An interview will be arranged where the subjects will be assessed for gastro-oesophageal symptoms using the Montreal GORD consensus definition and dysphagia based on the Hospital Odynophagia Dysphagia Questionnaire. Once confirmed asymptomatic, participants will be offered an appointment for enrolment. If candidates are asymptomatic, the subjects will be invited to a further interview where the procedure, risks and benefits will be discussed in detail. If participants fulfil the inclusion and exclusion criteria then participants will be given the option to enrol in the study. If at any point, participants wish to withdraw from the study, they have the option to do so without explaining why.

Once recruited the following assessments and interventions will take place:

1. Endoscopy and Bravo capsule placement under conscious sedation. The procedure will be performed by a trained endoscopist in using Bravo delivery system and dealing with any complications that may arise. Photographic documentation of capsule attachment will be taken.
2. 96-hour pH monitoring. Study subjects will be asked to document food intake, periods of sleep and occurrence of symptoms in a diary. After 96 hours, participants will return to the Oesophageal Laboratory to hand back in the receivers and diaries. The data captured on the recorder during the procedure will be downloaded to a computer.
3. Subjects will be offered a questionnaire detailing participants satisfaction with the overall study and an assessment of discomfort and interference with activities of daily living (diet, activity level) using a 5-point grading scale (1 = very unhappy/intolerant, 5 = very satisfied). A yes/no evaluation of participants ability to go to work or study on the day following the procedure and whether the participants would recommend this test to another person is also included.
4. Data analysis will include the standard components of oesophageal pH monitoring - acid exposure, number and duration of reflux episodes over 96 hours and 72 hours.
5. Statistical analysis will involve standard deviation, mean, median, 95th/5th percentiles and 25th/75th percentiles. Considering a 30% drop-out rate (the participants who cannot complete the test or their data is not useful), we will recruit 50 subjects to achieve 35

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic in:

  * GORD according to the Montreal GORD consensus definition
  * Dysphagia using the Hospital Odynophagia Dysphagia Questionnaire (HODQ) scoring < 7
* People without reflux referred for gastroscopy in context of other conditions e.g. iron deficiency anaemia, coeliac disease.
* Subjects must sign an informed consent

Exclusion Criteria:

* Gastro-oesophageal symptoms in accordance with Montreal criteria
* Previous abdominal operations on GI tract
* Antireflux treatments either prescribed or over the counter
* BMI > 35
* History of hepatic diseases, oesophageal varices
* History of ischemic heart disease, asthma
* Anticoagulants
* Allergies
* Pregnancy
* Any medical or non-medical condition that in the opinion of the research team will make the candidate unfit for this study e.g. drug abuse etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Acid exposure time in 4 days/96 hours | 4 days

SECONDARY OUTCOMES:
Acid exposure time in 3 days/72 hours | 3 days
Percent total time pH < 4 for each 24-hour period | 1 day
  Acid exposure measured as percent total time pH < 4
Percent Upright time pH < 4 for each 24-hour period | 1 day
  Acid exposure measured as percent Upright time pH < 4
Percent Supine time pH < 4 for each 24-hour period | 1 day
  Acid exposure measured as percent Supine time pH < 4
Number of reflux episodes for each 24-hour period | 1 day
  Acid exposure measured as number of reflux episodes
Number of reflux episodes ≥ 5 min for each 24-hour period | 1 day
  Acid exposure measured as number of reflux episodes ≥ 5 min
Longest reflux episode (minutes) for each 24-hour period | 1 day
  Acid exposure measured as the longest reflux episode (minutes)
Bravo "cut off" value for each 24-hour period | 1 day
  Acid exposure measured as Bravo "cut off" value

CONTACTS AND LOCATIONS:
Overall Officials: Terry Wong, MA MD, Principal Investigator — Consultant Gastroenterologist, Guy's and St Thomas' NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No